CLINICAL TRIAL: NCT07043010
Title: WHITE CAP Trial: Optical Parathyroid Tissue Sensor-Guided Assessment of Parathyroid Viability and Its Impact on Clinical Decision-Making
Brief Title: WHITE CAP: Intra-operative Parathyroid Tissue Sensor (PTS)-Guided Assessment of Parathyroid Viability and Surgical Decision-Making
Acronym: WHITE CAP-PTS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Bo Wang,MD, Director & Head of Thyroid Surgery, Principal Investigator, Clinical Professor, Fujian Medical University Union Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WHITECAP-PTS
Record Dates: First submitted 2025-06-21; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Hyperparathyroidism, Primary; Parathyroid Neoplasms; Parathyroid Adenoma; Hypocalcemia
Keywords: Near-Infrared Autofluorescence; Parathyroid Tissue Sensor; Parathyroid Viability; Peri-adenoma Rim Preservation; Intra-operative Imaging; Calcium Homeostasis; PTS Camera
MeSH Terms: conditions — Hyperparathyroidism, Primary; Parathyroid Neoplasms; Hypocalcemia

STUDY DESIGN:
Intervention Model Description: Randomized, parallel-group (1 : 1) controlled trial comparing preservation of peri-adenoma NIR-positive tissue with en-bloc excision.
Who Masked: Outcomes Assessor
Masking Description: Calcium and PTH assays will be processed and adjudicated by blinded laboratory personnel; investigators assessing primary endpoint are unaware of group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A - Rim Preservation (Experimental): Participants undergo adenoma removal guided by PTS imaging, with deliberate preservation of the NIR-autofluorescent rim of normal parathyroid tissue.
  Interventions: Device: Near-Infrared Parathyroid Tissue Sensor Imaging (PTS); Procedure: Rim-Preservation Technique
- Arm B - En-bloc Resection (Active Comparator): Participants undergo PTS-guided en-bloc excision of the adenoma plus its NIR-positive rim; parathyroid autotransplantation performed when indicated.
  Interventions: Device: Near-Infrared Parathyroid Tissue Sensor Imaging (PTS); Procedure: En-bloc Resection Technique

INTERVENTIONS:
Device: Near-Infrared Parathyroid Tissue Sensor Imaging (PTS) — FDA-cleared imager (e.g., Fluobeam LX/PTeye) providing real-time autofluorescence to identify parathyroid tissue during surgery; no dye or radiation.
Procedure: Rim-Preservation Technique — Surgical excision of adenoma while leaving the NIRAF-positive rim of normal parathyroid tissue in situ; minimal defatting to ensure perfusion.
  Arms: Arm A - Rim Preservation
Procedure: En-bloc Resection Technique — Surgical excision of adenoma together with the surrounding NIRAF-positive rim; autotransplant fragment if < 2 normal glands remain in neck.
  Arms: Arm B - En-bloc Resection

SUMMARY:
Primary hyperparathyroidism is usually cured by removing the single over-active parathyroid adenoma. During surgery, however, surgeons often see a thin rim of normal parathyroid tissue that still "glows" under a near-infrared parathyroid tissue sensor (PTS). It is unclear whether keeping this tissue in place helps preserve hormone function or whether it leaves behind cells that could become over-active again.

The WHITE CAP study will compare two common surgical choices:

Preservation strategy - the surgeon removes only the adenoma and leaves the glowing rim of normal tissue untouched.

En-bloc strategy - the surgeon removes the adenoma together with the glowing rim; if too little parathyroid tissue remains, a small fragment is transplanted into the forearm muscle.

About 120 adult patients who have a single parathyroid adenoma will be randomly assigned (like tossing a coin) to one of the two strategies. All operations will use the same FDA-cleared PTS camera that shows the glands in real time without dye or radiation.

The main question is whether preserving the normal rim lowers the rate of temporary low blood-calcium (numbness, tingling) during the first two days after surgery. The study will also check long-term results-blood calcium and parathyroid hormone (PTH) levels, symptoms, and any return of the disease-over two years.

The PTS imaging itself is painless and adds only a few minutes to the operation. Risks are the same as for standard parathyroid surgery, and participants can withdraw at any time without affecting their usual care.

DETAILED DESCRIPTION:
Background and Rationale Near-infrared autofluorescence (NIRAF) highlights parathyroid tissue at a wavelength of 820 nm. Several devices, including Fluobeam LX and PTeye®, have FDA 510(k) clearance for intra-operative identification of parathyroid glands. In ~70 % of single-gland disease, NIRAF shows a viable rim of normal tissue partially encasing the adenoma. Retrospective data conflict on whether rim preservation reduces transient hypocalcaemia or increases recurrence. No prospective randomized evidence exists.

Objectives Primary: Compare the incidence of transient hypocalcaemia (albumin-corrected Ca < 2.00 mmol·L-¹ or need for calcium/vit-D supplementation) within 48 h post-operative between preservation and en-bloc strategies.

Secondary: (i) Permanent hypocalcaemia at 6 months; (ii) PTH ≥ 15 pg·mL-¹ at 24 h; (iii) operative time and blood loss; (iv) biochemical or clinical recurrence up to 24 months; (v) correlation of quantitative NIRAF intensity with gland viability.

Study Design Multicentre, parallel-group, 1:1 randomized controlled trial (RCT). Block randomisation (size 4) stratified by centre and baseline vitamin-D status. Total sample 120 participants (60 per arm, includes 10 % attrition). Single-blind: outcome assessors and laboratory staff remain unaware of allocation.

Interventions Preservation arm: After adenoma excision, surgeon confirms NIRAF-positive rim and leaves it in situ; only minimal defatting to ensure vascularity.

En-bloc arm: Adenoma plus NIRAF-positive rim excised en bloc. If fewer than two normal glands remain in the neck, a 30 mg fragment is minced and autotransplanted into the non-dominant brachioradialis.

Eligibility Inclusion: age 18-75 y; biochemically confirmed primary hyperparathyroidism; imaging (MIBI or 4D-CT) concordant with a solitary adenoma; written informed consent.

Exclusion: multiple endocrine neoplasia, >1 enlarged gland on imaging, eGFR < 30, pregnancy, neck re-exploration, planned concomitant total thyroidectomy.

Outcome Assessments Serum Ca, phosphate, Mg, PTH measured pre-op; 6 h, 24 h, 48 h; Day 7; Months 1, 6, 12, 24. Laryngoscopy if voice change occurs. Recurrence defined as Ca above upper limit plus PTH > 65 pg·mL-¹ after Month 12. NIRAF intensity recorded (arbitrary units) using standard ROI software.

Statistical Plan Transient hypocalcaemia expected 30 % in en-bloc vs 10 % in preservation. With α = 0.05, 1-β = 0.80, needs 54 per arm; rounded to 60. Intent-to-treat analysis. Risk ratios with 95 % CI; secondary continuous outcomes by mixed-effects ANCOVA. Interim safety review at 50 % recruitment (O'Brien-Fleming boundary).

Regulatory and Ethics PTS devices are FDA-cleared; study classified as non-significant-risk device research exempt from IDE (21 CFR 812.2(b)). All centres have IRB approval. Data stored in REDCap, anonymised, GDPR-compliant. A three-member DSMB (endocrine surgeon, endocrinologist, biostatistician) will monitor AEs; trial pause if permanent hypocalcaemia exceeds 15 %.

Data Sharing De-identified participant data and analytic code will be available upon reasonable request 6 months after primary publication.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 75 years, able to give informed consent.
* Biochemically proven primary hyperparathyroidism (elevated serum calcium and inappropriately high PTH).
* Pre-operative imaging (sestamibi scan, 4-phase CT, or ultrasound) concordant with a single parathyroid adenoma.
* Planned minimally invasive parathyroidectomy using near-infrared parathyroid tissue sensor (PTS) guidance.

Exclusion Criteria:

* Multiple endocrine neoplasia (MEN 1 or 2) or suspicion of multi-gland disease (>1 enlarged gland on imaging).
* Prior parathyroid or extensive neck surgery causing distorted anatomy.
* Need for simultaneous total thyroidectomy or other major neck procedure.
* Estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m².
* Pregnancy or breastfeeding.
* Inability to tolerate general anaesthesia or contraindication to intra-operative PTS imaging.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Transient Hypocalcaemia | Baseline to 48 hours after surgery (Post-op Day 0-2)
  Proportion of participants whose albumin-corrected serum calcium falls < 2.00 mmol/L or who require oral/IV calcium ± active vitamin D to maintain normocalcaemia within 48 h post-operatively. Blood samples at 6 h, 24 h, and 48 h will be analysed by a blinded central laboratory.

SECONDARY OUTCOMES:
Permanent Hypocalcaemia | 6 months (±14 days) post-op
  Need for ongoing calcium ± calcitriol to maintain normocalcaemia at ≥ 6 months after surgery.
Parathyroid Hormone (PTH) Recovery ≥ 15 pg/mL | 24 hours post-op
  Percentage of patients with serum PTH ≥ 15 pg/mL at 24 h, indicating preserved parathyroid function.
Operative Time | Intra-operative (minutes)
  Skin incision to skin closure, recorded by anaesthesia time stamp.
Estimated Blood Loss | Intra-operative (mL)
  Calculated from suction canister minus irrigation plus soaked swab weight.
Biochemical or Clinical Recurrence | 12 to 24 months post-op
  Recurrence defined as serum calcium above lab upper limit of normal + PTH > 65 pg/mL and/or imaging-confirmed adenoma regrowth.
Correlation of NIRAF Intensity with PTH Recovery | Intra-op & 24 hours post-op
  Spearman correlation between quantitative NIRAF counts (ROI) and 24-h PTH value.

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided